CLINICAL TRIAL: NCT00974857
Title: Effects Of Volume Control Guided By Bioimpedance Spectroscopy On Blood Pressure And Cardiac Condition In Hemodialysis Patients
Brief Title: Effects Of Volume Control Guided by Body Composition Monitor (BCM) on Blood Pressure and Cardiac Condition in Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: Fresenius Medical Care North America (Industry)
Responsible Party: Principal Investigator, Ercan OK, Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 09-4/13
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Left Ventricular Hypertrophy
Keywords: Hemodialysis; Left Ventricular Hypertrophy; Body Composition Monitor
MeSH Terms: conditions — Hypertrophy, Left Ventricular | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study group (Active Comparator): Pre-dialytic overhydration(OH) will be estimated by Body Composition Monitor (BCM) at least once a month.
  1. If OH is positive, dry weight will be reached by ultrafiltration without regard to the level of blood pressure.
  2. If OH is negative and:
     * Systolic blood pressure(SBP)< 100 mmHg with/or intradialytic hypotension episodes(IDHE) and/or clothing and/or erythrocytosis(htc>36%);dry weight will be increased.
     * SBP normal(100-150 mmHg) w/o IDHE and clothing and erythrocytosis;dry weight will not be changed.
     * SBP normal(100-150 mmHg) with IDHE and/or clothing and/or erythrocytosis;dry weight will be increased.
     * SBP>150 mmHg captopril test(CT)will be done. If CT is positive, ACEI/ ARBs will be used and dry weight will be increased if IDHE and/or clothing and/or erythrocytosis(htc>36%) are present.
  If CT is negative, BCM measurement will be repeated and if same,ABPM will be performed for confirmation.
  Interventions: Device: BCM
- Control Group (Other): BCM results obtained at the beginning, at the 6th, and 12th months will not be given to the treating physicians. Dry weight estimation will be guided by clinical findings, telecardiography, and echocardiography as used to be.
  Interventions: Other: control group

INTERVENTIONS:
Device: BCM — Overhydration (OH) in liters will be estimated with the BCM (Body Composition Monitor, Fresenius Medical Care, Deutschland GmbH) in order to determine dry weight at least once a month before a dialysis session.
  Other Names: Body Composition Monitor,Fresenius Medical Care,Deutschland
  Arms: Study group
Other: control group — BCM results obtained at the beginning, at the 6th, and 12th months will not be given to the treating physicians. Dry weight estimation will be guided by clinical findings, telecardiography, and echocardiography as used to be.
  Arms: Control Group

SUMMARY:
This prospective, randomized, controlled study aims to evaluate the usefulness of the new body composition monitor (BCM) device as a method to improve volume control in hemodialysis (HD) patients and compare the results with those obtained by conventional volume control modalities.

DETAILED DESCRIPTION:
The proposed prospective, randomized, controlled study intends to document the effect of volume control guided by BCM on blood pressure (determined both manually and 48-h ambulatory), need for anti-hypertensive medication, intra-dialytic complications, and left ventricular geometry and functions assessed by echocardiography. One hundred and seventy-six prevalent HD patients will be randomized into two arms: study group and control group.

In the study group, "overhydration (OH) in liters" will be estimated with the BCM (Body Composition Monitor, Fresenius Medical Care, Deutschland GmbH)at least once a month before a dialysis session in order to determine dry weight.

1. If OH is positive value, we will try to reach dry weight by ultrafiltration without regard to the level of blood pressure.
2. If OH is negative value , and:

   * Systolic blood pressure is < 100 mmHg with/or intradialytic hypotension episodes and/or clothing and/or erythrocytosis ( htc> 36 %); we will increase dry weight accordingly.
   * Systolic blood pressure is normal (100-150 mmHg) without intradialytic hypotension episodes and clothing and erythrocytosis; we will not change dry weight.
   * Systolic blood pressure normal (100-150 mmHg) with intradialytic hypotension episodes and/or clothing and/or erythrocytosis; we will increase dry weight.
   * Systolic blood pressure> 150 mmHg we will perform a captopril test (CT) If the CT is positive we will use ACE inhibitors / ARBs as anti hypertensive drugs and dry weight will be increased if intradialytic hypotension episodes and/or clothing and/or erythrocytosis ( htc> 36 %) are also present

If the CT is negative we will repeat the BCM measurement and if it gives same results we will perform ABPM for confirmation.

We will not need to reach the dry weight immediately. If severe BP drop precludes reaching DW in one session, an isolated ultrafiltration or additional dialysis session will be added.

In the control group, BCM results obtained at the beginning, at the 6th, and 12th months will not be given to the treating physicians. Dry weight estimation will be guided by clinical findings, telecardiography, and echocardiography as used to be.

The planned duration of the study is 12 months. All patients will be seen in every month during the study. Additional visits will be scheduled if any symptoms and intolerance are suspected.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18-year,
* Maintenance bicarbonate HD scheduled thrice weekly (12 hours/week),
* Willingness to participate in the study with a written informed consent.

Exclusion Criteria:

* Presence of a cardiac stent, pacemaker or defibrillator ,
* Artificial joints, pin or amputation
* Permanent or temporary catheters (may affect BCM measurement),
* Being scheduled for living donor renal transplantation,
* Presence of serious life-limiting co-morbid situations, like malignancy, uncontrollable infection, end-stage cardiac, pulmonary, or hepatic disease,
* Pregnancy or lactating,
* Current use of investigational drugs or participation in an interventional clinical trial that contradicts or interferes with the therapies or measured outcomes in this trial,
* Mental incompetence.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Regression of left ventricular mass index (LVMI) | 1 year

SECONDARY OUTCOMES:
Changes in post-dialysis body weight | 1 year
Achievement of normal blood pressure level without using anti-hypertensive medication | 1 year
Decrease in left atrial volume | 1 year
Hematocrit and related rHu-EPO doses | 1 year
Serum levels of albumin and Hs-CRP | 1 year
Plasma level of pro-BNP | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ercan Ok, MD, Study Director — Ege University Division of Nephrology; Gulay Asci, MD, Principal Investigator — Ege University Division of Nephrology; Ender Hur, MD, Principal Investigator — Ege University Division of Nephrology
Locations (1):
- Ege University Division of Nephrology, Bornova, İzmir, Turkey (Türkiye)